CLINICAL TRIAL: NCT04570423
Title: A Multicenter, Open-Label, Phase 2 Study to Evaluate the Safety and Pharmacokinetics of Eflapegrastim in Pediatric Patients With Solid Tumors or Lymphomas and Treated With Myelosuppressive Chemotherapy
Brief Title: A Study to Evaluate the Safety and Pharmacokinetics of Eflapegrastim in Pediatric Participants With Solid Tumors or Lymphomas and Treated With Myelosuppressive Chemotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPI-GCF-202
Record Dates: First submitted 2020-09-15; First posted 2020-09-30 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumors; Lymphoma
Keywords: Lymphomas; Solid Tumors; Chemotherapy
MeSH Terms: conditions — Lymphoma | interventions — eflapegrastim; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: ≥12 to <17 years (Experimental): Participants will receive a SC injection of eflapegrastim after completion of each cycle of chemotherapy up to four cycles of treatment (cycle length may vary and can be up to 28 days or more based on the type of chemotherapy regimen selected).
  Interventions: Drug: Eflapegrastim; Drug: Chemotherapy
- Cohort 2: ≥6 to <12 years (Experimental): Participants will receive a SC injection eflapegrastim after completion of each cycle of chemotherapy up to four cycles of treatment (cycle length may vary and can be up to 28 days or more based on the type of chemotherapy regimen selected).
  Interventions: Drug: Eflapegrastim; Drug: Chemotherapy
- Cohort 3: ≥2 to <6 years (Experimental): Participants will receive a SC injection eflapegrastim after completion of each cycle of chemotherapy up to four cycles of treatment (cycle length may vary and can be up to 28 days or more based on the type of chemotherapy regimen selected).
  Interventions: Drug: Eflapegrastim; Drug: Chemotherapy
- Cohort 4: ≥1 month to <2 years (Experimental): Participants will receive a SC injection eflapegrastim after completion of each cycle of chemotherapy up to four cycles of treatment (cycle length may vary and can be up to 28 days or more based on the type of chemotherapy regimen selected).
  Interventions: Drug: Eflapegrastim; Drug: Chemotherapy

INTERVENTIONS:
Drug: Eflapegrastim — Eflapegrastim supplied in prefilled, single-use syringes for SC injection.
  Other Names: Rolontis®; SPI-2012
Drug: Chemotherapy — Chemotherapy agents may include doxorubicin, ifosfamide, docetaxel, CHOP regimen, etoposide, cyclophosphamide and vincristine which will be administered as per standard of care per the Primary Care physician's treatment plan.

SUMMARY:
The purpose of this study is to evaluate the safety and pharmacokinetics of eflapegrastim in pediatric participants with solid tumors or lymphoma and treated with myelosuppressive chemotherapy.

DETAILED DESCRIPTION:
This is a Phase 2, open label, multicenter study of eflapegrastim in pediatric participants (≥1 month to <17 years) with solid tumors or lymphoma.

Approximately 40 participants will be enrolled and assigned to one of 4 age-based cohorts. Participants enrolled in Cohort 1 will be followed for dose-limiting toxicities (DLTs) prior to initiating parallel enrollment into Cohorts 2 through 4.

All participants will receive chemotherapy as Standard of Care after which a subcutaneous (SC) dose of eflapegrastim will be administered up to 4 treatment cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must have a pathologic/histologic confirmed newly diagnosed/relapsed/recurrent solid tumor or lymphoma without bone marrow involvement.
2. Participant must be a candidate to receive myelosuppressive chemotherapy, with a febrile neutropenia rate of at least 20% as outlined in the National Comprehensive Cancer Network (NCCN) guidelines.
3. Participant has adequate hematological, renal, and hepatic function.
4. Participant must have an echocardiogram (ECHO) or multigated acquisition (MUGA) within 14 days of Screening if receiving a cardiotoxic therapy and have a cardiac ejection fraction of >50%.
5. Participant must have a lumbar puncture, if clinically indicated, to rule out central nervous system (CNS) involvement within 14 days of study entry.
6. Participant has a Karnofsky performance level ≥50% for patients ≥16 years of age or a Lansky performance level ≥50 for children <16 years of age.

Exclusion Criteria:

1. Participant has an uncontrollable infection, has an underlying medical condition, and/or another serious illness that would impair the ability of the participant to receive protocol-specified treatment.
2. Participant has had previous exposure to filgrastim (within 7 days), pegfilgrastim (within 14 days), or other granulocyte colony stimulating factor (G-CSF) products in clinical development within 2 weeks prior to the administration of study drug (eflapegrastim)
3. Participant requires concurrent radiation therapy specifically in Cycle 1.
4. Participant has had prior bone marrow or hematopoietic stem cell transplant and/or has concurrent bone marrow involvement in their malignancy, including leukemia.
5. Participant has had spinal radiation therapy within 30 days prior to study enrollment.
6. Participant has used any investigational drugs, biologics or devices within 30 days prior to study treatment or plans to use any of these during the study.
7. Participant has a known sensitivity or previous reactions to any of the G-CSF products.
8. Participant with active CNS disease.
9. Participant has not recovered from previous treatment adverse events to ≤Grade 1.

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events (TEAEs) | From first dose of study drug to 35 days after the last dose of the study drug (Up to approximately 16 months)
  An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A TEAE is any AE that occurs from the first dose of the study drug until 35 days after the last dose of study drug, or on the day a new/additional chemotherapy regimen, or on the day another granulocyte-colony stimulating factor (G-CSF) is administered.

SECONDARY OUTCOMES:
Percentage of Participants With Severe Neutropenia in Cycle 1 | Cycle 1 (cycle length may vary and can be up to 28 days or more based on the type of chemotherapy selected)
  Severe neutropenia is defined as absolute neutrophil count (ANC) less than 0.5*10^9/liter (L).
Time to Absolute Neutrophil Count (ANC) Recovery of Severe Neutropenia in Cycle 1 | Cycle 1 (cycle length may vary and can be up to 28 days or more based on the type of chemotherapy selected)
  Time to ANC recovery of severe neutropenia is defined as the time from chemotherapy administration until the participants ANC increases to ≥1.0*10^9/L after the expected nadir.
Number of Participants With Febrile Neutropenia in Cycle 1 | Cycle 1 (cycle length may vary and can be up to 28 days or more based on the type of chemotherapy selected)
  Febrile neutropenia is defined as ANC less than 0.5*10^9/L with a single temperature of >38.3 degree Celsius (°C) or a sustained temperature of ≥38°C for more than 1 hour.
Peak Concentration (Cmax) of Eflapegrastim in Cycle 1 | Pre-dose and at multiple time points (up to Day 9 [Cohorts 1-3] and Day 6 [Cohort 4]) post-dose in Cycle 1 (cycle length may vary and can be up to 28 days or more based on the type of chemotherapy selected)
Time to Reach Peak Concentration (Tmax) of Eflapegrastim in Cycle 1 | Pre-dose and at multiple time points (up to Day 9 [Cohorts 1-3] and Day 6 [Cohort 4]) post-dose in Cycle 1 (cycle length may vary and can be up to 28 days or more based on the type of chemotherapy selected)
Elimination Half-life (t½) of Eflapegrastim in Cycle 1 | Pre-dose and at multiple time points (up to Day 9 [Cohorts 1-3] and Day 6 [Cohort 4]) post-dose in Cycle 1 (cycle length may vary and can be up to 28 days or more based on the type of chemotherapy selected)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - New York Medical College, Valhalla, New York
  - Carolinas Medical Center/ Levine Children's Hospital, Charlotte, North Carolina
  - Levine Children's Health, Charlotte, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - UT MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No